CLINICAL TRIAL: NCT00237367
Title: A Randomized, Two-way Crossover Study of the Effects of a Single Dose of Rabeprazole or Pantoprazole on 24-hour Intragastric Acidity and Esophageal Acid Exposure in GERD Patients With a History of Nocturnal Heartburn
Brief Title: A Study of Rabeprazole and Pantoprazole on Stomach Acid and Esophageal Acid Exposure in Patients With Gastroesophageal Reflux Disease (GERD) and a History of Nighttime Heartburn
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Collaborators: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR004618
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; GERD; Nighttime heartburn; heartburn; esophagus; esophageal acid exposure; EAE; Aciphex; Pariet; rabeprazole; Protonix; pantoprazole
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Rabeprazole; Pantoprazole

INTERVENTIONS:
Drug: rabeprazole and pantoprazole

SUMMARY:
The purpose of the study is to compare the pharmacodynamics (the way a drug works in the body) of rabeprazole and pantoprazole on intragastric acidity and esophageal acid exposure in gastroesophageal reflux disease (GERD) patients with nighttime heartburn. Patients will be given one dose of each medication with a washout period of 6 to 13 days between doses ("washout period" means they will receive no further proton pump inhibitor medication for 6-13 days, allowing the 1st dose to completely leave their bodies). Rabeprazole is approved in the United States for the short-term treatment (4-8 weeks) in the healing and symptomatic relief of erosive or ulcerative GERD with symptoms of daytime or nighttime heartburn, maintenance of healing of erosive or ulcerative GERD, and treatment of symptomatic GERD. The dosage regimen for all GERD indications is 20 mg once a day. Other indications include healing of duodenal ulcers, Helicobacter pylori eradication to reduce the risk of duodenal ulcer recurrence, and treatment of pathological hypersecretory conditions including Zollinger-Ellison Syndrome. The most common side effect of rabeprazole is headache. In clinical trials headache was assessed as possibly related to rabeprazole in 2.4% of subjects vs. 1.6% for placebo. Pantoprazole at a dose of 40 mg once a day is indicated for the short-term treatment (up to 8 weeks) in the healing and symptomatic relief of erosive esophagitis, and the maintenance of healing of erosive esophagitis and reduction in relapse rates of daytime and nighttime heartburn symptoms in patients with GERD. Other indications include pathological hypersecretory conditions including Zollinger-Ellison Syndrome. The most common side effects are headache and diarrhea.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effects of a single dose of two drugs, rabeprazole and pantoprazole, on reducing the amount of acid in the stomach and esophagus in subjects with GERD. This study is conducted at one investigational center. The investigator will be blinded (he or she will not know whether the patient is taking rabeprazole or pantoprazole). The study is a comparative, randomized, single dose, two-way crossover, pharmacodynamic study examining the effectiveness of rabeprazole or pantoprazole on stomach acidity and esophageal acid exposure in GERD patients with nighttime heartburn. Patients will be randomized (like with the toss of a coin) to one of two sequences in receiving study medication; either one dose of rabeprazole in the first treatment period followed by one dose of pantoprazole in the second treatment period or one dose of pantoprazole in the first treatment period followed by one dose of rabeprazole in the second treatment period. The study will measure how the acid levels in the stomach and esophagus change after one dose of either study medication. The primary endpoint will be the percent of time that the stomach pH is greater than 4 (a pH level considered to be normal) during the 24-hour period after a single dose of each study medication. Another endpoint will be the 24-hour esophageal reflux time after a single dose of study medication. The esophageal acid exposure is determined by measuring how much acid flows backwards from the stomach to the esophagus. Patients will participate in two 48-hour treatment periods during which intragastric (stomach) and esophageal pH will be recorded at 8-second intervals using a probe inserted through the nose and down to the stomach. The two treatment periods will be be separated by a washout period of 6 to 13 days. On each day of the treatment periods, patients will be dosed in the morning. During each treatment period, patients will receive placebo on Day 1, and active treatment (either rabeprazole or pantoprazole) on Day 2. The main objective of the study is to compare the effects of a single dose of rabeprazole 20 milligrams to pantoprazole 40 milligrams on intragastric acidity and esophageal acid exposure in GERD patients with a history of nighttime heartburn and safety will be monitored in the study. Rabeprazole 20 milligram tablet once by mouth; pantoprazole 40 milligram tablet once by mouth

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GERD with symptoms for at least 6 months with at least 3 episodes a week and one of those at nighttime
* in generally good health
* stop any previous similar (proton pump inhibitor) therapy at least 10 days before screening
* weigh within normal weight for one's height
* able to tolerate a nasogastric tube (pH probe assembly that goes through the nose into the stomach) for 48 hours on 2 different occasions
* esophageal acid exposure of at least 10% on a 24-hour pH monitoring study performed within the 24 months prior to screening
* Helicobacter pylori (an infection) negative
* willing to take only TUMS antacid as rescue medicine during the washout period

Exclusion Criteria:

* History of a serious medical condition
* significant gastrointestinal illness other than GERD
* ulcer at any time in the past
* difficulty swallowing
* history of gastrointestinal disease (including bleeding)
* use of any medication that changes acid secretion or gastrointestinal movement in the past 14 days
* use of any drugs on a list of prohibited drugs within 1 month
* chronic use of pain relieving medications (NSAIDs or COX-2 inhibitors)
* pregnant or breast-feeding
* cancer diagnosis or treatment (except for superficial skin cancers)
* abusing drugs or alcohol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics: intragastric pH measurements, collected every 8 seconds for each 24 hour period after administration of study medication on Day 1 and Day 2 of each study period; percent of the 24-hour period with intragastric pH>4

SECONDARY OUTCOMES:
Pharmacodynamics: esophageal pH measurements, collected every 8 seconds for each 24 hour period after administration of study drug on Day 1 and Day 2 of each study period; 24-hour esophageal acid reflex time (percent 24-hour period with esophageal pH<4)

CONTACTS AND LOCATIONS:
Overall Officials: PriCara, Unit of Ortho-McNeil, Inc. Clinical Trial, Study Director — PriCara, Unit of Ortho-McNeil, Inc.

REFERENCES:
- [Derived] Miner P, Delemos B, Xiang J, Lococo J, Ieni J. Effects of a single dose of rabeprazole 20 mg and pantoprazole 40 mg on 24-h intragastric acidity and oesophageal acid exposure: a randomized study in gastro-oesophageal reflux disease patients with a history of nocturnal heartburn. Aliment Pharmacol Ther. 2010 May;31(9):991-1000. doi: 10.1111/j.1365-2036.2010.04255.x. Epub 2010 Feb 2. PMID 20132153